CLINICAL TRIAL: NCT00207376
Title: Prospective Multicenter Clinical Study to Evaluate the Safety and Effectiveness of an Intracardiac Septal Closure Device in Patients With Atrial Septum Defect (ASD) and Patent Foramen Ovale (PFO)
Brief Title: Safety and Effectiveness Study of the Solysafe Septal Occluder in Patients With Atrial Septum Defect and Patent Foramen Ovale
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Carag AG (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 04k001
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2009-06-24 (Estimated); Status verified 2007-02

CONDITIONS: Atrial Septal Defect; Patent Foramen Ovale
MeSH Terms: conditions — Heart Septal Defects, Atrial; Foramen Ovale, Patent

INTERVENTIONS:
Device: Solysafe Septal Occluder

SUMMARY:
This is a prospective multicenter clinical study to evaluate the safety and effectiveness of an intracardiac septal closure device in patients with atrial septum defect (ASD) and patent foramen ovale (PFO).

ELIGIBILITY:
Inclusion Criteria:

* ASD
* PFO with a medical history of cryptogenic stroke due to presumed paradoxical embolism caused by a PFO

Exclusion Criteria:

* Criteria that exclude catheterization (e.g. size too small, disseminated intravascular coagulopathy (DIC), high risk of bleeding such as coagulation or clotting disorders)

Min Age: 3 Years | Sex: All
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Peter Ewert, PD Dr., Principal Investigator — German Heart Institute
Locations (1):
- German Heart Institute, Berlin, Germany